CLINICAL TRIAL: NCT02312323
Title: One-month Clinical Evaluation of Silicone Hydrogel Definitive 65 HPT Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contamac Ltd (Industry)
Collaborators: Hartwig Research Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM-001-002
Record Dates: First submitted 2014-11-28; First posted 2014-12-09 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

ARMS (2):
- Definitive 65 HPT (Experimental): The Test product were the Definitive 65 (Filcon V4) lenses with Hydra PEG surface coating. This material is produced by Contamac Ltd. and the contact lenses were manufactured by Appenzeller Kontaktlinsen AG.
  Interventions: Device: Definitive 65 HPT contact lenses
- Definitive 65 (Active Comparator): The Control product was the commercially available Definitive 65 (Efrofilcon A) lens. This material is produced by Contamac Ltd. and the contact lenses were manufactured by Appenzeller Kontaktlinsen AG.
  Interventions: Device: Definitive 65 contact lenses

INTERVENTIONS:
Device: Definitive 65 HPT contact lenses
  Other Names: Filcon V4 (HPT)
  Arms: Definitive 65 HPT
Device: Definitive 65 contact lenses
  Other Names: Filcon V4
  Arms: Definitive 65

SUMMARY:
Comparison of different contact lens materials.

DETAILED DESCRIPTION:
This is a 1-month, open-label, bilateral, parallel-group, randomised, daily wear study. Two-thirds of the subjects will wear the Test lenses in both eyes, and one-third will wear the Control lenses in both eyes.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to sign informed consent form
* ages 18 years or older
* Subjects must have owned spectacles or contact lenses prior to enrolment for this trial
* Spherical power between -10.00 D and +10.00 D (at vertex distance 0 mm)
* Astigmatic power ≤0.75 D

Exclusion Criteria:

* Eye injury or surgery within 3 months immediately prior to enrolment for this trial
* Pre-existing ocular irritation that would preclude contact lens fitting
* Currently enrolled in an ophthalmic clinical trial
* Evidence of systemic or ocular abnormality, infection or disease which is likely to affect successful wear of contact lenses or use of the accessory solutions, as determined by the investigator
* Any use of medications for which contact lens wear could be contradicted, as determined by the investigator
* Current extended-wear users (sleep-in overnight)
* Current monovision lens wearers
* Pregnant women and nursing mothers
* Best-corrected visual acuity worse than 6/9 (LogMAR: +0.20; Snellen decimal: 0.63)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-11-08 (Actual); Primary Completion 2015-05-23 (Actual); Study Completion 2015-05-23 (Actual)

PRIMARY OUTCOMES:
questionnaire addressing subjective comfort and wear time | subjects will be followed-up for one month
  Subjects rated on a scale from 1 to 10, where 1 was 'poor' and 10 was 'excellent'.
limbal redness - ocular biomicroscopy | subjects will be followed-up for one month
  Assessed using slit lamp with white light, low-medium magnification. Graded based on a grading scale which ranged from 0 to 4, where 0 is none, 1 is trace, 2 is mild, 3 is moderate and 4 is severe.
conjunctival redness - ocular biomicroscopy | subjects will be followed-up for one month
  Assessed using slit lamp with white light, low-medium magnification. Graded based on a grading scale which ranged from 0 to 4, where 0 is none, 1 is trace, 2 is mild, 3 is moderate and 4 is severe.
corneal staining - ocular biomicroscopy | subjects will be followed-up for one month
  Assessed using slit lamp with white light, low-medium magnification. Graded based on a grading scale which ranged from 0 to 4, where 0 is none, 1 is trace, 2 is mild, 3 is moderate and 4 is severe.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hartwig, PhD, FAAO, Principal Investigator — Hartwig Research Center
Locations (2):
- Germany (2):
  - Siehste, Kassel
  - Kresinky, Würzburg